CLINICAL TRIAL: NCT01071694
Title: QOLBET Quality Of Life in Patients With Early Relapsing-remitting Multiple Sclerosis Treated With BETaferon® in Korea
Status: Withdrawn | Type: Observational
Why Stopped: Study Manager could not embark on it during the timeline.
Sponsor: Bayer (Industry)
Responsible Party: Global Medical Affairs Therapeutic area Head, Bayer HealthCare AG
Other Study IDs: 15110; Qolbet (Other: Company internal); BF1010KR (Other: Company internal)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis,; Relapsing-Remitting,; Interferon beta-1b,; Quality of life
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta 1-b (Betaferon/Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta 1-b (Betaferon/Betaseron, BAY86-5046) — Patients receiving Betaferon according to routine clinical practice

SUMMARY:
This study is to describe the quality of life of Korean patients with early relapsing-remitting multiple sclerosis during the initial 1 year of treatment with Betaferon with several validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS (RRMS) patients within the first two years after diagnosis according to Poser or McDonald criteria, starting Betaferon treatment, including patients switching from other DMDs
* Patients who signed informed consent form

Exclusion Criteria:

* Age lower than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life evaluated by several validated questionnaire | Baseline, 3, 6, 9, 12 months (+/- 1 month)

SECONDARY OUTCOMES:
Information about safety of Betaferon in routine clinical use | Baseline, 3, 6, 9, 12 months (+/- 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea